CLINICAL TRIAL: NCT05138653
Title: A Phase 1, Double-blind (Investigator and Participant), First-in-Human Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of CVL-354 in Healthy Participants
Brief Title: A Single and Multiple Ascending Dose Trial of CVL-354 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerevel Therapeutics, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CVL-354-1001; 1UG3DA052166-01A1 (NIH)
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Healthy Participants
Keywords: Healthy Volunteer; CVL-354

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (15):
- Part A: Cohort 1: Sequence 1 (Experimental): Participants were randomized to sequence 1 to receive placebo on Day 1 of Period 1 followed by CVL-354 1.5 milligrams (mg) on Day 1 of Period 2, followed by CVL-354 5 mg on Day 1 of Period 3 & followed by CVL-354 15 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 1: Sequence 2 (Experimental): Participants were randomized to sequence 2 to receive CVL-354 0.5 mg on Day 1 of Period 1 followed by placebo on Day 1 of Period 2, followed by CVL-354 5 mg on Day 1 of Period 3 & followed by CVL-354 15 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 1: Sequence 3 (Experimental): Participants were randomized to sequence 3 to receive CVL-354 0.5 mg on Day 1 of Period 1 followed by CVL-354 1.5 mg on Day 1 of Period 2, followed by placebo on Day 1 of Period 3 & followed by CVL-354 15 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 1: Sequence 4 (Experimental): Participants were randomized to sequence 4 to receive CVL-354 0.5 mg on Day 1 of Period 1 followed by CVL-354 1.5 mg on Day 1 of Period 2, followed by CVL-354 5 mg on Day 1 of Period 3 & followed by placebo on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 2: Sequence 1 (Experimental): Participants were randomized to sequence 1 to receive placebo on Day 1 of Period 1 followed by CVL-354 90 mg on Day 1 of Period 2, followed by CVL-354 150 mg on Day 1 of Period 3 & followed by CVL-354 200 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 2: Sequence 2 (Experimental): Participants were randomized to sequence 2 to receive CVL-354 45 mg on Day 1 of Period 1 followed by placebo on Day 1 of Period 2, followed by CVL-354 150 mg on Day 1 of Period 3 & followed by CVL-354 200 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 2: Sequence 3 (Experimental): Participants were randomized to sequence 3 to receive CVL-354 45 mg on Day 1 of Period 1 followed by CVL-354 on 90 mg Day 1 of Period 2, followed by placebo on Day 1 of Period 3 & followed by CVL-354 200 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 2: Sequence 4 (Experimental): Participants were randomized to sequence 4 to receive CVL-354 45 mg on Day 1 of Period 1 followed by CVL-354 90 mg on Day 1 of Period 2, followed by CVL-354 150 mg on Day 1 of Period 3 & placebo on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part A: Cohort 3: Sequence 1: Fed/Fasted Sequence (Experimental): Participants first received a single oral dose of CVL-354 50 mg, under fed state on Day 1 of Period 1 followed by a single oral dose of CVL-354 50 mg under fasted state on Day 1 of Period 2, with a washout period of 2 days between both periods.
  Interventions: Drug: CVL-354
- Part A: Cohort 3: Sequence 2: Fasted/Fed Sequence (Experimental): Participants first received a single oral dose of CVL-354 50 mg, under fasted state on Day 1 of Period 1 followed by a single oral dose of CVL-354 50 mg under fed state on Day 1 of Period 2, with a washout period of 2 days between both periods
  Interventions: Drug: CVL-354
- Part B: Cohort 1: CVL-354 10 mg (Experimental): Participants received oral dose of CVL-354 10 mg or Placebo, once daily (QD) from Day 1 up to Day 14 in Cohort 1.
  Interventions: Drug: CVL-354; Drug: Placebo
- Part B: Cohort 2: CVL-354 25 mg (Experimental): Participants received oral dose of CVL-354 25 mg or Placebo, QD from Day 1 up to Day 14 in Cohort 2.
  Interventions: Drug: Placebo; Drug: CVL-354
- Part B: Cohort 3: CVL-354 50 mg (Experimental): Participants received oral dose of CVL-354 50 mg or Placebo, QD from Day 1 up to Day 14 in Cohort 3.
  Interventions: Drug: Placebo; Drug: CVL-354
- Part B: Cohort 4: CVL-354 80 mg (Experimental): Participants received oral dose of CVL-354 80 mg or Placebo, QD from Day 1 up to Day 14 in Cohort 4.
  Interventions: Drug: Placebo; Drug: CVL-354
- Part B: Cohort 5: CVL-354 85 mg (Experimental): Participants received oral dose of CVL-354 85 mg or Placebo, QD from Day 1 up to Day 14 in Cohort 5.
  Interventions: Drug: Placebo; Drug: CVL-354

INTERVENTIONS:
Drug: CVL-354 — Oral solution/suspension
  Arms: Part A: Cohort 1: Sequence 1; Part A: Cohort 1: Sequence 2; Part A: Cohort 1: Sequence 3; Part A: Cohort 1: Sequence 4; Part A: Cohort 2: Sequence 1; Part A: Cohort 2: Sequence 2; Part A: Cohort 2: Sequence 3; Part A: Cohort 2: Sequence 4; Part B: Cohort 1: CVL-354 10 mg
Drug: Placebo — Placebo matched to CVL-354
  Arms: Part A: Cohort 1: Sequence 1; Part A: Cohort 1: Sequence 2; Part A: Cohort 1: Sequence 3; Part A: Cohort 1: Sequence 4; Part A: Cohort 2: Sequence 1; Part A: Cohort 2: Sequence 2; Part A: Cohort 2: Sequence 3; Part A: Cohort 2: Sequence 4; Part B: Cohort 1: CVL-354 10 mg; Part B: Cohort 2: CVL-354 25 mg; Part B: Cohort 3: CVL-354 50 mg; Part B: Cohort 4: CVL-354 80 mg; Part B: Cohort 5: CVL-354 85 mg
Drug: CVL-354 — Capsule
  Arms: Part A: Cohort 3: Sequence 1: Fed/Fasted Sequence; Part A: Cohort 3: Sequence 2: Fasted/Fed Sequence; Part B: Cohort 2: CVL-354 25 mg; Part B: Cohort 3: CVL-354 50 mg; Part B: Cohort 4: CVL-354 80 mg; Part B: Cohort 5: CVL-354 85 mg

SUMMARY:
This is a 2-part, double-blind, randomized, placebo-controlled, first-in-human trial evaluating a single ascending dose (4-way crossover, Part A) and multiple ascending doses (Part B) of CVL-354.

ELIGIBILITY:
Inclusion Criteria:

1. Women of nonchildbearing potential and men 18 to 55 years, inclusive.
2. Healthy as determined by medical evaluation, including medical and psychiatric history, physical and neurological examinations, Electrocardiogram (ECG), vital sign measurements, and laboratory test results, as evaluated by the investigator.
3. Body mass index of 18.5 to 30.0 Kilograms per square meter (kg/m^2), inclusive, and total body weight >50 Kilogram (kg) [110 Pound (lb)] at Screening.
4. A male participant with a pregnant or a nonpregnant partner of childbearing potential must agree to use contraception during the trial and 14 days following the last dose of study drug.
5. Capable of giving signed informed consent
6. Ability, in the opinion of the investigator, to understand the nature of the trial and comply with protocol requirements.

Exclusion Criteria:

1. Current or past history of significant cardiovascular, pulmonary, gastrointestinal, renal, hepatic, metabolic, genitourinary, endocrine, hematological, immunological, or neurological, or psychiatric disease that, in the opinion of the investigator or medical monitor, could compromise either participant safety or the results of the trial.
2. Serious risk of suicide in the opinion of the Investigator
3. History of substance or alcohol-use disorder (excluding nicotine or caffeine) within 12 months prior to signing the informed consent form (ICF).
4. Any condition that could possibly affect drug absorption
5. Receipt of severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccination or booster as follows:

   * messenger ribonucleic acid (mRNA): within 14 days prior to dosing
   * Non-mRNA: within 28 days prior to dosing In addition, participants who plan to receive SARS-CoV2 vaccination or booster while participating in the trial or for at least 14 days after the last dose of investigational medicinal product (IMP) will be excluded.
6. Have recently been diagnosed with symptomatic corona virus disease-2019 (COVID-19) or test positive for COVID-19 within 30 days prior to signing the ICF.
7. Use of prohibited medication prior to randomization or likely to require prohibited concomitant therapy (eg, prescription and over-the-counter medications, herbal medications, vitamins, and supplements) during the trial
8. Either of the following:

   * History of human immunodeficiency viruses (HIV), hepatitis B, or hepatitis C infection
   * Positive result for HIV antibody, hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C antibody
9. Positive drug screen (including nicotine) or a positive test for alcohol
10. Abnormal clinical laboratory test results or vital measurements at Screening and Check-in
11. Estimated glomerular filtration rate at Screening <90 millilitre/minute/1.73m^2 (mL/min/1.73 m^2), as calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
12. Abnormal 12-lead ECG at Screening or initial Check-In (Day -1).
13. Known allergy or hypersensitivity to the IMP, closely related compounds, or any of their specified ingredients.
14. Current enrollment or past participation within 30 days or 5 half-lives (whichever is longer) prior to signing the ICF in any other clinical trial involving an IMP.
15. Any other abnormal safety findings unless, based on the investigator's judgment, the findings are not medically significant and would not impact the safety of the participant or the interpretation of the trial results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, MD, MBA, Study Director — Cerevel Therapeutics, LLC
Locations (1):
- Labcorp Drug Development, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 participants took part in the study at 1 investigative site in the United States of America from 18 October 2021 to 23 January 2023.
Pre-assignment Details: Healthy participants were enrolled in single ascending dose (Part A: Cohorts 1 & 2), food effect (Part A: Cohorts 3) & multiple ascending dose (Part B: Cohorts 1-5) of the study. The data for the 4 sequences in Cohorts 1 and 2 was collected and presented in a pooled manner in the participant flow.
Groups:
- Part A: Cohort 2: Sequence 4: Participants were randomized to sequence 4 to receive CVL- 354 45 mg on Day 1 of Period 1 followed by CVL-354 90 mg on Day 1 of Period 2, followed by CVL-354 150 mg on Day 1 of Period 3 & placebo on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
- Part A: Cohort 3: Fed/Fasted Sequence: Participants first received a single oral dose of CVL-354 50 mg, under fed state on Day 1 of Period 1 followed by a single oral dose of CVL-354 50 mg under fasted state on Day 1 of Period 2, with a washout period of 2 days between both periods.
- Part A: Cohort 3: Fasted/Fed Sequence: Participants first received a single oral dose of CVL-354 50 mg, under fasted state on Day 1 of Period 1 followed by a single oral dose of CVL-354 50 mg under fed state on Day 1 of Period 2, with a washout period of 2 days between both periods.
- Part B: Pooled Placebo: Participants received oral dose of placebo matching CVL-354, once daily (QD) from Day 1 up to Day 14 of Cohort 1 to 5 in Part B.
- Part B: Cohort 1: CVL-354 10 mg: Participants received oral dose of CVL-354 10 mg, QD from Day 1 up to Day 14 in Cohort 1.
- Part B: Cohort 2: CVL-354 25 mg: Participants received oral dose of CVL-354 25 mg, QD from Day 1 up to Day 14 in Cohort 2.
- Part B: Cohort 3: CVL-354 50 mg: Participants received oral dose of CVL-354 50 mg, QD from Day 1 up to Day 14 in Cohort 3.
- Part B: Cohort 4: CVL-354 80 mg: Participants received oral dose of CVL-354 80 mg, QD from Day 1 up to Day 14 in Cohort 4.
- Part B: Cohort 5: CVL-354 85 mg: Participants received oral dose of CVL-354 85 mg, QD from Day 1 up to Day 14 in Cohort 5.
Period: Single Ascending Dose (Up to 13 Weeks)
Arm/Group | Part A: Cohort 1: Sequence 1 | Part A: Cohort 1: Sequence 2 | Part A: Cohort 1: Sequence 3 | Part A: Cohort 1: Sequence 4 | Part A: Cohort 2: Sequence 1 | Part A: Cohort 2: Sequence 2 | Part A: Cohort 2: Sequence 3 | Part A: Cohort 2: Sequence 4 | Part A: Cohort 3: Fed/Fasted Sequence | Part A: Cohort 3: Fasted/Fed Sequence | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Started | 2 | 4 | 2 | 2 | 3 | 2 | 3 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Investigator's Discretion | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Multiple Ascending Dose (Up to 12 Weeks)
Arm/Group | Part A: Cohort 1: Sequence 1 | Part A: Cohort 1: Sequence 2 | Part A: Cohort 1: Sequence 3 | Part A: Cohort 1: Sequence 4 | Part A: Cohort 2: Sequence 1 | Part A: Cohort 2: Sequence 2 | Part A: Cohort 2: Sequence 3 | Part A: Cohort 2: Sequence 4 | Part A: Cohort 3: Fed/Fasted Sequence | Part A: Cohort 3: Fasted/Fed Sequence | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 8 | 6 | 7 | 8 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8 | 5 | 6 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disciplinary Reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Population included all participants who were randomized to investigational medicinal product (IMP).
Groups:
- Part A: Cohort 1: Sequence 1: Participants were randomized to sequence 1 to receive placebo on Day 1 of Period 1 followed by CVL-354 1.5 mg on Day 1 of Period 2, followed by CVL-354 5 mg on Day 1 of Period 3 & followed by CVL-354 15 mg on Day 1 of Period 4. Each dosing period was separated by a washout period of at least 5 days.
- Part B: Pooled Placebo: Participants received oral dose of placebo matching CVL-354, QD from Day 1 up to Day 14 of Cohort 1 to 5 in Part B.
- Total: Total of all reporting groups
Arm/Group | Part A: Cohort 1: Sequence 1 | Part A: Cohort 1: Sequence 2 | Part A: Cohort 1: Sequence 3 | Part A: Cohort 1: Sequence 4 | Part A: Cohort 2: Sequence 1 | Part A: Cohort 2: Sequence 2 | Part A: Cohort 2: Sequence 3 | Part A: Cohort 2: Sequence 4 | Part A: Cohort 3: Fed/Fasted Sequence | Part A: Cohort 3: Fasted/Fed Sequence | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg | Total
Number analyzed (Participants) | 2 | 4 | 2 | 2 | 3 | 2 | 3 | 2 | 4 | 3 | 9 | 8 | 6 | 7 | 8 | 8 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 2 | 2 | 3 | 2 | 3 | 2 | 4 | 3 | 9 | 8 | 6 | 7 | 8 | 8 | 73
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 6
  Male | 2 | 3 | 2 | 2 | 2 | 2 | 3 | 2 | 3 | 2 | 8 | 8 | 6 | 7 | 8 | 7 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 0 | 3 | 2 | 1 | 19
  Not Hispanic or Latino | 2 | 4 | 1 | 2 | 0 | 2 | 2 | 0 | 3 | 2 | 8 | 5 | 6 | 4 | 6 | 7 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 0 | 7 | 4 | 5 | 2 | 5 | 4 | 38
  White | 0 | 1 | 1 | 0 | 3 | 1 | 2 | 1 | 2 | 2 | 2 | 3 | 1 | 4 | 3 | 2 | 28
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Cohorts 1 and 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of trial treatment, whether or not considered related to the trial treatment. A serious adverse event (SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Adverse event which was reported to have started on Day 1 with no associated onset time were defined as TEAEs. TEAEs included both serious and non-serious TEAEs.
Time Frame: From the first dose of study drug up to end of follow-up period (Up to 72 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 1 and 2: Pooled Placebo: Participants received a single oral dose of placebo matching CVL-354 on Day 1 of either of the 4 periods in Cohorts 1 and 2 of Part A.
- Part A: Cohort 1: CVL-354 0.5 mg: Participants received a single oral dose of CVL-354 0.5 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 1: CVL-354 1.5 mg: Participants received a single oral dose of CVL-354 1.5 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 1: CVL-354 5 mg: Participants received a single oral dose of CVL-354 5 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 1: CVL-354 15 mg: Participants received a single oral dose of CVL-354 15 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 2: CVL-354 45 mg: Participants received a single oral dose of CVL-354 45 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 2: CVL-354 90 mg: Participants received a single oral dose of CVL-354 90 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 2: CVL-354 150 mg: Participants received a single oral dose of CVL-354 150 mg on Day 1 of either of the 4 periods.
- Part A: Cohort 2: CVL-354 200 mg: Participants received a single oral dose of CVL-354 200 mg on Day 1 of either of the 4 periods.
Arm/Group | Part A: Cohort 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 5 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 2

2. Primary Outcome: Part A: Cohorts 1 and 2: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: ECG parameters were assessed using continuous ECG recordings and standard 12-lead ECGs. The parameters included heart rhythm, heart rate, QRS intervals, QT intervals, RR intervals, PR intervals, corrected QT (QTc) intervals, corrected QT with Bazett formula (QTcB), and corrected QT with Fredericia (QTcF) parameters measurement. Clinical significance of changes in ECG parameters was based on investigator's interpretation. Number of participants with clinically significant changes in ECG were reported.
Time Frame: From the first dose of study drug up to end of treatment (Up to 72 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 5 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part A: Cohorts 1 and 2: Number of Participants With Clinically Significant Changes in Vital Sign Measurements
Description: Vital signs include systolic and diastolic blood pressures, heart rate, respiratory rate, and body temperature. Clinical significance of changes in vital signs measurements was based on investigator's interpretation. Number of participants with clinically significant changes in vital signs were reported.
Time Frame: From the first dose of study drug up to end of treatment (Up to 72 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 5 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part A: Cohorts 1 and 2: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: Laboratory parameters included blood chemistry, hematology, and urinalysis. Clinical significance of changes in laboratory parameters was based on investigator's interpretation. Number of participants with clinically significant changes in laboratory parameters (included hematology, blood chemistry, and urinalysis) were reported.
Time Frame: From the first dose of study drug up to end of treatment (Up to 72 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 5 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part A: Cohorts 1 and 2: Number of Participants With Clinically Significant Changes in Physical and Neurological Examinations
Description: The full physical examination included a review of the following body systems: head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, and musculoskeletal systems. The full neurological examination included an assessment of the participant's mental status (level of consciousness, orientation, speech, memory, etc), cranial nerves, motor (muscle appearance, tone, strength and reflexes), sensation (including Romberg sign), coordination, and gait. Clinical significance in changes of physical and neurological examination results were based on investigator's interpretation. Number of participants with clinically significant changes in physical and neurological examinations were reported.
Time Frame: From the first dose of study drug up to end of treatment (Up to 72 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 5 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Part A: Cohorts 1 and 2: Number of Participants With Changes in Suicidal Ideation or Suicidal Behavior Assessed Using the Columbia Suicide-Severity Rating Scale (C-SSRS)
Description: The C-SSRS is comprised of 10 categories with binary responses. The 10 categories include: Category 1 - Wish to be Dead; Category 2 - Non-specific Active Suicidal Thoughts; Category 3 - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Category 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Category 5 - Active Suicidal Ideation with Specific Plan and Intent; Category 6 - Preparatory Acts or Behavior; Category 7 - Aborted Attempt; Category 8 - Interrupted Attempt; Category 9 - Actual Attempt (non-fatal); Category 10 - Completed Suicide. Categories 1-5 represent Suicidal Ideation and categories 6-10 represent Suicidal Behavior. Each category is scored as 1 if there is a positive response in the category and a 0 if there are no positive responses in the category.
Time Frame: From the first dose of study drug up to end of treatment (Up to 72 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 5 | 5 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Part A: Cohort 3: Number of Participants With TEAEs
Description: An AE was any untoward medical occurrence in a clinical trial participant, temporally associated with the use of trial treatment, whether or not considered related to the trial treatment. A SAE was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Adverse event which was reported to have started on Day 1 with no associated onset time were defined as TEAEs. TEAEs included both serious and non-serious TEAEs.
Time Frame: From the first dose of study drug up to end of follow up period (Up to 22 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 3: Fed State: Participants received a single oral dose of CVL-354 50 mg under fed state on Day 1 of either Period 1 or Period 2.
- Part A: Cohort 3: Fasted State: Participants received a single oral dose of CVL-354 50 mg under fasted state on Day 1 of either Period 1 or Period 2.
Arm/Group | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted State
Number analyzed (Participants) | 7 | 7
Participants | 0 | 2

8. Primary Outcome: Part A: Cohorts 3: Number of Participants With Clinically Significant Changes in ECG Parameters
Description: as for outcome 2
Time Frame: From the first dose of study drug up to end of treatment (Up to 22 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted State
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

9. Primary Outcome: Part A: Cohorts 3: Number of Participants With Clinically Significant Changes in Vital Sign Measurements
Description: as for outcome 3
Time Frame: From the first dose of study drug up to end of treatment (Up to 22 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted State
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

10. Primary Outcome: Part A: Cohorts 3: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: as for outcome 4
Time Frame: From the first dose of study drug up to end of treatment (Up to 22 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted State
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

11. Primary Outcome: Part A: Cohort 3: Number of Participants With Clinically Significant Changes in Physical and Neurological Examinations
Description: as for outcome 5
Time Frame: From the first dose of study drug up to end of treatment (Up to 22 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 3: Fasted State: Participants received a single oral dose of CVL-354 50 mg under fasted state on Day 1 either of Period 1 or Period 2.
Arm/Group | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted State
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

12. Primary Outcome: Part A: Cohort 3: Number of Participants With Changes in C-SSRS
Description: as for outcome 6
Time Frame: From the first dose of study drug up to end of treatment (Up to 22 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part A: Cohort 3: Fasted Stated: Participants received a single oral dose of CVL-354 50 mg under fasted state on Day 1 of either Period 1 or Period 2.
Arm/Group | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted Stated
Number analyzed (Participants) | 7 | 7
Participants | 0 | 0

13. Primary Outcome: Part B: Number of Participants With TEAEs
Description: as for outcome 7
Time Frame: From the first dose of study drug up to end of follow up period (Up to 31 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Cohort 2: CVL-354 25 mg: Participants received oral doses of CVL-354 25 mg, QD from Day 1 up to Day 14 in Cohort 2.
- Part B: Cohort 3: CVL-354 50 mg: Participants received oral doses of CVL-354 50 mg, QD from Day 1 up to Day 14 in Cohort 3.
- Part B: Cohort 4: CVL-354 80 mg: Participants received oral doses of CVL-354 80 mg, QD from Day 1 up to Day 14 in Cohort 4.
- Part B: Cohort 5: CVL-354 85 mg: Participants received oral doses of CVL-354 85 mg, QD from Day 1 up to Day 14 in Cohort 5.
Arm/Group | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Number analyzed (Participants) | 9 | 8 | 6 | 7 | 8 | 8
Participants | 2 | 0 | 1 | 2 | 2 | 3

14. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in ECG Parameters
Description: as for outcome 2
Time Frame: From the first dose of study drug up to end of treatment (Up to 31 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Number analyzed (Participants) | 9 | 8 | 6 | 7 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

15. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Vital Sign Measurements
Description: as for outcome 3
Time Frame: From the first dose of study drug up to end of treatment (Up to 31 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Cohort 2: CVL-354 50 mg: Participants received oral doses of CVL-354 50 mg, QD from Day 1 up to Day 14 in Cohort 3.
- Part B: Cohort 3: CVL-354 80 mg: Participants received oral doses of CVL-354 80 mg, QD from Day 1 up to Day 14 in Cohort 4.
Arm/Group | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 2: CVL-354 50 mg | Part B: Cohort 3: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Number analyzed (Participants) | 9 | 8 | 6 | 7 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

16. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Clinical Laboratory Parameters
Description: as for outcome 4
Time Frame: From the first dose of study drug up to end of treatment (Up to 31 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Number analyzed (Participants) | 9 | 8 | 6 | 7 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

17. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Physical and Neurological Examinations
Description: as for outcome 5
Time Frame: From the first dose of study drug up to end of treatment (Up to 31 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Number analyzed (Participants) | 9 | 8 | 6 | 7 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Part B: Number of Participants With Changes in C-SSRS
Description: The C-SSRS is comprised of 10 categories with binary responses. The 10 categories include: Category 1 - Wish to be Dead; Category 2 - Non-specific Active Suicidal Thoughts; Category 3 - Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Category 4 - Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Category 5 - Active Suicidal Ideation with Specific Plan and Intent; Category 6 - Preparatory Acts or Behavior; Category 7 - Aborted Attempt; Category 8 - Interrupted Attempt; Category 9 - Actual Attempt (non-fatal); Category 10 - Completed Suicide. Categories 1-5 represent Suicidal Ideation and categories 6-10 represent Suicidal Behavior Each category is scored as 1 if there is a positive response in the category and a 0 if there are no positive responses in the category.
Time Frame: From the first dose of study drug up to end of treatment (Up to 31 days)
Population: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
Number analyzed (Participants) | 9 | 8 | 6 | 7 | 8 | 8
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A: Cohorts 1 and 2: From the first dose of study drug up to end of follow up period (Up to 72 days); Part A: Cohort 3: From the first dose of study drug up to end of follow up period (Up to 22 days); Part B: From the first dose of study drug up to end of follow up period (Up to 31 days)
Description: Safety Analysis Set included all randomized participants who had received at least 1 dose of IMP.
Groups:
- Part A: Cohorts 1 and 2: Pooled Placebo: Participants received a single oral dose of placebo matching CVL-354 on Day 1 of either of the 4 periods in Cohorts 1 and 2 of Part A.
Arm/Group | Part A: Cohorts 1 and 2: Pooled Placebo | Part A: Cohort 1: CVL-354 0.5 mg | Part A: Cohort 1: CVL-354 1.5 mg | Part A: Cohort 1: CVL-354 5 mg | Part A: Cohort 1: CVL-354 15 mg | Part A: Cohort 2: CVL-354 45 mg | Part A: Cohort 2: CVL-354 90 mg | Part A: Cohort 2: CVL-354 150 mg | Part A: Cohort 2: CVL-354 200 mg | Part A: Cohort 3: Fed State | Part A: Cohort 3: Fasted State | Part B: Pooled Placebo | Part B: Cohort 1: CVL-354 10 mg | Part B: Cohort 2: CVL-354 25 mg | Part B: Cohort 3: CVL-354 50 mg | Part B: Cohort 4: CVL-354 80 mg | Part B: Cohort 5: CVL-354 85 mg
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/4 | 0/6 | 0/6 | 0/7 | 0/7 | 0/9 | 0/8 | 0/6 | 0/7 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/5 | 0/5 | 0/4 | 0/6 | 0/6 | 0/7 | 0/7 | 0/9 | 0/8 | 0/6 | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 1/6 | 0/5 | 1/5 | 0/4 | 2/6 | 2/6 | 0/7 | 2/7 | 2/9 | 0/8 | 1/6 | 2/7 | 2/8 | 3/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Cohorts 1 and 2: Pooled Placebo (N=16) | Part A: Cohort 1: CVL-354 0.5 mg (N=6) | Part A: Cohort 1: CVL-354 1.5 mg (N=6) | Part A: Cohort 1: CVL-354 5 mg (N=6) | Part A: Cohort 1: CVL-354 15 mg (N=5) | Part A: Cohort 2: CVL-354 45 mg (N=5) | Part A: Cohort 2: CVL-354 90 mg (N=4) | Part A: Cohort 2: CVL-354 150 mg (N=6) | Part A: Cohort 2: CVL-354 200 mg (N=6) | Part A: Cohort 3: Fed State (N=7) | Part A: Cohort 3: Fasted State (N=7) | Part B: Pooled Placebo (N=9) | Part B: Cohort 1: CVL-354 10 mg (N=8) | Part B: Cohort 2: CVL-354 25 mg (N=6) | Part B: Cohort 3: CVL-354 50 mg (N=7) | Part B: Cohort 4: CVL-354 80 mg (N=8) | Part B: Cohort 5: CVL-354 85 mg (N=8)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronavirus disease 2019 (COVID-19) (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Product taste abnormal (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urethritis chlamydial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-05-25): https://cdn.clinicaltrials.gov/large-docs/53/NCT05138653/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-17): https://cdn.clinicaltrials.gov/large-docs/53/NCT05138653/SAP_001.pdf